CLINICAL TRIAL: NCT06956716
Title: Clinical Study to Evaluate the Safety and Efficacy of Personalized Tumor Neoantigen mRNA Therapy in Combination With PD-1 Antibody and Chemotherapy for Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Personalized Tumor Neoantigen mRNA Therapy for Advanced Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-14
Record Dates: First submitted 2025-04-09; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Advanced Intrahepatic Cholangiocarcinoma
MeSH Terms: interventions — Gemcitabine; Cisplatin; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Experimental)
  Interventions: Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection; Drug: Gemcitabine + cisplatin (GP); Drug: Sintilimab injection

INTERVENTIONS:
Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection — The individualized anti-tumor new antigen iNeo-Vac-R01 injection was commissioned by Hangzhou Nuanjin Biotechnology Co., Ltd., and all patients were admitted into the therapeutic intervention group. According to the results of previous non-clinical studies, the individualized mRNA injection of 100 μ g was a tolerable dose.
Drug: Gemcitabine + cisplatin (GP) — As standard chemotherapy (D1, D8 gemcitabine 1000mg/m², intravenous drip for 30 minutes, cisplatin 25mg/m², intravenous drip), once every 3 weeks
Drug: Sintilimab injection — Sintilimab Injection, 200mg, intravenous infusion

SUMMARY:
The main purpose of this study is to evaluate the feasibility and safety of personalized tumor neoantigen mRNA therapy iNeo-Vac-R01 combined with PD-1 monoclonal antibody and standard chemotherapy regimen for the treatment of patients with advanced intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects who meet all the following inclusion criteria will enter the pre-screening stage of this study and undergo the lesion puncture process:

  1. Voluntarily sign the informed consent form;
  2. Aged ≥18 years and ≤75 years, regardless of gender;
  3. Imaging assessment of unresectable advanced intrahepatic cholangiocarcinoma;
  4. Have not received systemic or local treatment.
  5. According to the solid tumor efficacy evaluation criteria (RECIST 1.1), the investigators assess the lesions as measurable.
  6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
  7. Adequate fresh tumor tissue samples can be obtained for exome and transcriptome sequencing analysis;
  8. Normal function of the main organs of the heart, liver and kidney:

     1. QTc (corrected QT interval) in the electrocardiogram: ≤450 milliseconds for men, or ≤470 milliseconds for women;
     2. Coagulation function: international normalized ratio (INR) ≤1.5×ULN; activated partial thromboplastin time (APTT) ≤1.5 times ULN;
     3. Hematological indicators: white blood cells ≥3.5×109/L; absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin (HGB) ≥10 g/dL; platelet count (PLT) ≥80×109/L;
     4. Biochemical indicators: serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN (ALT or AST ≤ 5 times ULN is allowed for patients with liver metastasis and liver cancer); serum creatinine and urea nitrogen ≤ 1.5 times ULN;
  9. Male and female patients of childbearing age with fertility agree to take effective contraceptive measures from the signing of the informed consent form to 6 months after the last dose of the trial drug; women of childbearing age include premenopausal women and women within 2 years after menopause;
  10. Able to follow the study protocol and follow-up procedures.

  (2) Subjects who meet all the following inclusion criteria will enter the formal screening stage of this study and enter the study medication process:
  1. Voluntary signing of the informed consent form;
  2. Age ≥ 18 years and ≤ 75 years, regardless of gender;
  3. Intrahepatic cholangiocarcinoma confirmed by pathology (histology or cytology);
  4. Have not received any systemic treatment.
  5. According to the solid tumor efficacy evaluation criteria (RECIST 1.1), the investigators assessed the patients as having measurable lesions.
  6. The Eastern Cooperative Oncology Group (ECOG) performance status score was 0 or 1;
  7. The major organ functions of the heart, liver, and kidney were normal:

     1. QTc (corrected QT interval) in the electrocardiogram: ≤450 milliseconds for men or ≤470 milliseconds for women;
     2. Coagulation function: international normalized ratio (INR) ≤1.5×ULN; activated partial thromboplastin time (APTT) ≤1.5 times ULN;
     3. Hematological indicators: white blood cells ≥3.5×109/L; absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin (HGB) ≥10 g/dL; platelet count (PLT) ≥80×109/L;
     4. Biochemical indicators: serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN (ALT or AST ≤ 5 times ULN is allowed for patients with liver metastasis and liver cancer); serum creatinine and urea nitrogen ≤ 1.5 times ULN;
  8. Male patients with fertility and female patients of childbearing age agree to take effective contraceptive measures from the signing of the informed consent form to 6 months after the last administration of the trial drug; women of childbearing age include premenopausal women and women within 2 years after menopause;
  9. Able to follow the study protocol and follow-up process.

     Exclusion Criteria:
* If the subject meets any of the following criteria, he/she will be excluded from this study:

  1. Those who suffer from other malignant tumors at the same time, but have been cured of basal cell carcinoma, thyroid cancer, cervical atypical hyperplasia, etc., have been in a disease-free state for more than 5 years or are considered by the researchers to be less likely to relapse;
  2. Those who have received a history of bone marrow transplantation, allogeneic organ transplantation, or allogeneic hematopoietic stem cell transplantation;
  3. Those who are accompanied by immunosuppressants, that is, those who need to take immunosuppressants regularly 4 weeks before the screening period and during the clinical study, including but not limited to the following situations: those with severe asthma, autoimmune diseases or immunodeficiency, those who are treated with immunosuppressive drugs, and those with a known history of primary immunodeficiency; but type 1 diabetes, autoimmune-related hypothyroidism requiring hormone treatment, and vitiligo and psoriasis that do not require systemic treatment are excluded;
  4. Active bacterial or fungal infection confirmed by clinical diagnosis; active tuberculosis or history of tuberculosis;
  5. Positive test results for human immunodeficiency virus (HIV) antibody, positive test results for Treponema pallidum (TP), active hepatitis C (positive hepatitis C virus (HCV) antibody and positive HCV RNA), active hepatitis B;
  6. Herpes virus infection (except for those with scabs for more than 4 weeks); respiratory virus infection (except for those who have recovered for more than 4 weeks);
  7. Uncontrolled complications include but are not limited to active infection, symptomatic congestive heart failure, unstable angina, arrhythmia; severe coronary artery disease or cerebrovascular disease, or other diseases that the investigator considers unsuitable for inclusion;
  8. History of drug abuse, clinical, psychological or social factors that affect informed consent or research implementation; history of mental illness;
  9. History of food, drug or vaccine allergy, or other potential immunotherapy allergy considered by the investigator.
  10. Pregnant or lactating women;
  11. Those who the investigator considers unsuitable for inclusion or may not be able to complete this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerable dose | 21±3 days after the last dose
  According to the Commonly Used Adverse Events Criteria (CTCAE Version 5.0), the number of subjects with adverse events and/or dose-limiting toxicity was counted as an indicator of the safety and tolerable dose of iNeo-Vac-R01 injection. The evaluation period was the dosing observation period and the safety follow-up period.

SECONDARY OUTCOMES:
Objective reponse rate (ORR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR according to RECIST1.1 criteria during the whole study
Disease control rate (DCR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR or SD according to RECIST1.1 criteria during the whole study.
Progression-free survival （PFS） | Up to 2 years
  The time from enrolled to disease pregression or death from any cause during the whole study.
Overall survival (OS) | Up to 2 years
  The time from enrolled to death from any cause during the whole study.
Overall Survival Rate (1-Y-OS%,2-Y-OS%,3-Y-OS%) | Up to 3 years
  The percentage of patients surviving at 12, 24, and 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No